CLINICAL TRIAL: NCT01424865
Title: Evaluation of the Co-Expression of the Cancer Stem Cell Marker ALDH1 and of HER2 as a Predictor of Adjuvant Trastuzumab Response in Breast Cancers of Women in NSABP B31
Brief Title: Cancer Stem Cell Biomarkers as a Predictor of Response to Trastuzumab in Samples From Patients With Breast Cancer Previously Treated in the NSABP-B-31 Trial
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NSABP B-31 ICSCA; NSABP-B31-ICSC-A
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: HER2-positive breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — In Situ Hybridization, Fluorescence; Immunohistochemistry; Immunologic Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Other: immunohistochemistry staining method
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers as a predictor of response to trastuzumab in samples from patients with breast cancer previously treated in the NSABP-B-31 trial.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if stem cellness identifies a poor prognostic subgroup of women with early-stage breast cancer who have been uniformly treated with either adjuvant doxorubicin hydrochloride & cyclophosphamide followed by paclitaxel (the "control arm" of B31), or the same chemotherapy plus trastuzumab.

Secondary

* To conduct exploratory analyses to assess, to the extent possible, if co-localization of stem cellness, as determined by ALDH1 positivity, and HER2 identifies a group of patients previously considered to have HER2-negative cancers (using classical definitions) who benefit from adjuvant trastuzumab.

OUTLINE: Archived breast cancer stem cells samples and terminally differentiated cells from tissue samples are analyzed for HER2 and ALDH1 expression by dual-staining quantitative immunofluorescence using Automated Quantitative Analysis (AQUA) , IHC, and fluorescence in situ hybridization (FISH).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tissue samples from patients with node-positive breast cancer whose tumors overexpress HER2
* Primary tumor samples that are negative for HER2 using classically accepted cutoffs determined in the metastatic setting
* Treated with adjuvant therapy comprising doxorubicin hydrochloride, cyclophosphamide, and paclitaxel with or without trastuzumab in the NSABP-B-31 trial

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary cancer tissue from participants in protocol NSABP B-31.
Sampling Method: Non-Probability Sample
Enrollment: 1874 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
ALDH1 expression (percentage of stem cells within the tumor) and association with outcomes regardless of HER2 staining | approximately 4 years

SECONDARY OUTCOMES:
HER2 expression in cells with stem cell-like properties as a determinant of aggressiveness and response to trastuzumab in the adjuvant setting | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F. Hayes, MD, Principal Investigator — University of Michigan Rogel Cancer Center